CLINICAL TRIAL: NCT03230552
Title: Effect of Pre-operative Training Using Surgical Videos on Resident Performance of Unilateral Salpigo-oophrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17-124
Record Dates: First submitted 2017-07-24; First posted 2017-07-26 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Surgical Videos; Pre-operative Training

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video group (Experimental): Residents assigned to this group will watch an instructional surgical video prior to LSO surgery.
  Interventions: Other: Instructional surgical video
- No video group (No Intervention): Residents assigned to this group will not watch an instructional surgical video prior to LSO surgery.

INTERVENTIONS:
Other: Instructional surgical video — An instructional surgical video shown to residents before they perform LSO surgery.
  Arms: Video group

SUMMARY:
There is a need for the development and validation of new teaching strategies and resources for surgical training that can occur outside of the operating room. The use of surgical videos is not novel however it has not been validated as an effective approach for gynecologic surgical training. The goals of our study are to (1) develop an educational surgical video for laparoscopic salpingo-oophrectomy (LSO) and (2) to evaluate and test the effectiveness of this tool in preparing residents for performance in the operating room.

DETAILED DESCRIPTION:
In the rapidly changing face of surgical education and with a pressure to adopt competency-based training and assessment nationwide, obstetrics and gynecology residency programs will be forced to implement effective strategies to ensure that learners acquire the skill set required to become competent gynecologists. However, very few instructional tools have been validated in gynecologic surgery. The use of surgical videos as a teaching strategy may be one piece to this puzzle. Surgical videos are becoming increasingly popular, however, their value as an effective instructional technique has yet to be validated. Should surgical videos prove to be of benefit in surgical training it would offer an alternate modality to optimize operating room experiences and learning for gynecology residents.

Obstetrics and gynecology residents in years one and two of their training (junior residents), will view a teaching video about LSO (intervention group) compared to not watching a video (control group) to assess if our intervention results in better performance in the operating room for this procedure as rated by an objective structured assessment of technical skills tool (OSAT) (primary outcome). Secondary outcome measures will include a self-administered questionnaire grading knowledge and confidence, and a 5-point Likert scale grading resident satisfaction with the video.

ELIGIBILITY:
Inclusion Criteria:

* Novice OBGYN residents who have performed <10 LSO surgeries as the primary surgeon

Exclusion Criteria:

* OBGYN residents who have performed > 10 LSO surgeries as the primary surgeon.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
Objective Structure Assessment of Technical Skills Tool (OSAT) | Intraoperative (Beginning of surgery to end of surgery)
  Surgeries performed by the residents will be video recorded. Resident performance during surgery will be rated using the OSAT tool.

SECONDARY OUTCOMES:
Pre-operative knowledge survey | baseline
  Residents will complete a survey prior surgery which will measure their pre-operative knowledge of performing LSO procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Eliane Shore, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Norris S, Papillon-Smith J, Gagnon LH, Jacobson M, Sobel M, Shore EM. Effect of a Surgical Teaching Video on Resident Performance of a Laparoscopic Salpingo-oophorectomy: A Randomized Controlled Trial. J Minim Invasive Gynecol. 2020 Nov-Dec;27(7):1545-1551. doi: 10.1016/j.jmig.2020.01.010. Epub 2020 Jan 23. PMID 31982585